CLINICAL TRIAL: NCT00243035
Title: A Dose Escalation Study of R115777 (Zarnestra) Combined With Velcade® (PS-341) in Patients With Relapsed Multiple Myeloma.
Brief Title: Tipifarnib and Bortezomib in Treating Patients With Relapsed Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02675; NCI-2012-02675 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MCC-VEL-04-111; CDR0000446083; NCI-7032; VEL-04-111 (Other: H. Lee Moffitt Cancer Center and Research Institute); 7032 (Other: CTEP); R01CA083978 (NIH)
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Refractory Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; tipifarnib

ARMS (1):
- Treatment (bortezomib, tipifarnib) (Experimental): Phase I: Patients receive bortezomib IV on days 1, 4, 8, and 11 and oral tipifarnib twice daily on days 1-14. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of tipifarnib until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. An additional 6 patients are treated at the MTD.
  Phase II: Patients receive bortezomib as in phase I and tipifarnib as in phase I at the MTD.
  Interventions: Drug: bortezomib; Drug: tipifarnib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bortezomib — Given IV
Drug: tipifarnib — Given orally
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I/II trial is studying the side effects and best dose of tipifarnib when given together with bortezomib and to see how well they work in treating patients with relapsed multiple myeloma. Tipifarnib and bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving tipifarnib together with bortezomib may kill more cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES: Primary I. Determine the maximum tolerated dose and dose-limiting toxicity of tipifarnib when administered with bortezomib in patients with relapsed multiple myeloma. (Phase I) II. Determine the response rate in patients treated with this regimen. (Phase II) III. Determine the toxicity profile of this regimen in these patients. (Phase II)

Secondary I. Determine the progression-free survival of patients treated with this regimen. (Phase II)

Tertiary I. Determine whether this regimen overcomes CAM-DR in primary myeloma cells and establish whether ex vivo efficacy predicts a clinical response in these patients.

II. Determine if activated Akt predicts clinical resistance and if levels of phosphorylated Akt are reduced by tipifarnib and bortezomib in these patients.

III. Determine whether molecular profiles from primary isolates (suspension vs adhered) correlate with clinical response in patients treated with this regimen.

OUTLINE: This is a phase I dose-escalation study of tipifarnib followed by a phase II study.

Phase I: Patients receive bortezomib IV on days 1, 4, 8, and 11 and oral tipifarnib twice daily on days 1-14. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of tipifarnib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. An additional 6 patients are treated at the MTD.

Phase II: Patients receive bortezomib as in phase I and tipifarnib as in phase I at the MTD.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: Approximately 52-64 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma

  * Stage II or III disease
* Relapsed disease after ≥ 2 prior therapies*, confirmed by the presence of 1 of the following:

  * New lytic lesion
  * A 25% increase in urine or serum monoclonal protein
* Patients who received prior bortezomib must have responded to therapy
* Measurable disease, defined by 1 or more of the following criteria:

  * Serum M-component ≥ 1.0 g/dL by serum protein electrophoresis
  * Urine M-protein excretion > 200 mg per 24-hour collection, by urine protein electrophoresis
* Performance status - Karnofsky 60-100%
* More than 8 weeks
* Platelet count ≥ 100,000/mm^3
* Absolute neutrophil count ≥ 1,000/mm^3
* Bilirubin ≤ 2 mg/dL
* Direct bilirubin ≤ 2 times upper limit of normal (ULN)
* AST or ALT ≤ 2 times ULN
* Creatinine ≤ 1.5 times ULN
* Calcium ≤ 12 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow study medication
* Capable of following directions regarding study medication, or has a daily caregiver who will be responsible for administering study medication
* No peripheral neuropathy ≥ grade 2
* No hypersensitivity to any of the following:

  * Bortezomib
  * Boron
  * Mannitol
  * Imidazole compounds (e.g., clotrimazole, ketoconazole, miconazole, econazole)
* No serious medical or psychiatric illness that would preclude study compliance
* No other life-threatening illness (unrelated to tumor)
* No other active or invasive malignancy within the past 3 years except for nonmelanoma skin cancer
* No serious infection
* No prior allogeneic bone marrow transplantation
* More than 30 days since prior and no concurrent immunotherapy
* More than 30 days since prior and no concurrent cytotoxic chemotherapy
* More than 14 days since prior high-dose corticosteroids
* No concurrent therapeutic corticosteroids (e.g., > 10 mg prednisone per day)
* No concurrent hormonal therapy
* No concurrent antiemetic corticosteroids
* More than 14 days since prior and no concurrent radiotherapy
* More than 1 year since prior bortezomib
* More than 14 days since prior investigational drugs
* No prior tipifarnib
* No other concurrent cancer-related treatment
* No concurrent administration of the following enzyme-inducing anti-epileptic drugs:

  * Phenytoin
  * Phenobarbital
  * Carbamazepine
* No concurrent magnesium- or aluminum-based antacids within 2 hours before or after tipifarnib administration
* Concurrent pamidronate or other bisphosphonates allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2005-08; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of tipifarnib as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0 (phase I) | Up to day 21
Response rate (complete response [CR] + partial response [PR]) determined using the Bladé Response criteria (phase II) | Up to 6 weeks
  Exact 95% confidence intervals constructed.
Toxicities, graded according to the NCI CTCAE v3.0 (phase II) | Up to 2 years

SECONDARY OUTCOMES:
Proportion of patients overcoming CAM-DR | Prior to therapy
  An exact 95% confidence interval for that proportion will be computed.
Proportion of patients overcoming CAM-DR | Day 11 of course 1
  An exact 95% confidence interval for that proportion will be computed.
Relationship of overcoming CAM-DR and clinical response | Prior to therapy
  Compared using a chi-square contingency table test at the two-sided 0.05 significance level.
Relationship of overcoming CAM-DR and clinical response | Day 11 of course 1
  Compared using a chi-square contingency table test at the two-sided 0.05 significance level.
Clinical resistance and levels of phosphorylated Akt | Prior to therapy
  P-Akt levels both pre and post treatment will be obtained and compared using a paired t test. Logistic regression will be used with P-Akt activity as independent variable in a logistic regression modeling probability of response. Odds ratio indicating change in odds of response associated with a unit change in P-Akt level will be computed as well as a 95% confidence interval for that odds ratio.
Clinical resistance and levels of phosphorylated Akt | Day 11 of course 1
  P-Akt levels both pre and post treatment will be obtained and compared using a paired t test. Logistic regression will be used with P-Akt activity as independent variable in a logistic regression modeling probability of response. Odds ratio indicating change in odds of response associated with a unit change in P-Akt level will be computed as well as a 95% confidence interval for that odds ratio.
Correlation of molecular profiles from primary isolates with clinical response | Prior to therapy
  Compared using paired t tests at the 0.05 significance level.
Correlation of molecular profiles from primary isolates with clinical response | Day 11 of course 1
  Compared using paired t tests at the 0.05 significance level.
Progression-free survival (phase II) | Up to 2 years
  Summarized with Kaplan-Meier curve and related statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Darrin Beaupre, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States